CLINICAL TRIAL: NCT05243628
Title: ABC [Afrezza With Basal Combination]: A Phase 4 Study of Mealtime Control With Afrezza in Adult Subjects With Type 1 Diabetes Mellitus in Combination With an Automated Insulin Pump or Insulin Degludec
Brief Title: Afrezza With Basal Combination (ABC): Afrezza® Combined With AID Pump or Insulin Degludec in Adults With Type 1 Diabetes
Acronym: ABC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-192
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Mellitus; Insulin; Inhaled Insulin; Afrezza; Technosphere Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Insulin; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Afrezza + Automatic Insulin Delivery (Experimental): Subjects in this group will use Afrezza for their bolus (mealtime) insulin and a CSII pump with an AID algorithm using RAA for their basal and correction insulin coverage.
  Interventions: Biological: Afrezza (insulin human) Inhalation Powder; Device: Continuous Subcutaneous Insulin Infusion (CSII) pump with Automatic Insulin Delivery (AID)
- Afrezza + Insulin Degludec (Experimental): Subjects in this group will use Afrezza for their bolus (mealtime and correction) insulin and insulin degludec for basal insulin coverage.
  Interventions: Biological: Afrezza (insulin human) Inhalation Powder; Biological: insulin degludec
- AID Control (Active Comparator): Subjects in this group will use a CSII pump with an AID algorithm using RAA for all bolus (mealtime and correction) and basal insulin coverage (control group).
  Interventions: Device: Continuous Subcutaneous Insulin Infusion (CSII) pump with Automatic Insulin Delivery (AID)

INTERVENTIONS:
Biological: Afrezza (insulin human) Inhalation Powder — Pharmaceutical form: powder
  Route of administration: inhalation
  Other Names: Technosphere Insulin
  Arms: Afrezza + Automatic Insulin Delivery; Afrezza + Insulin Degludec
Biological: insulin degludec — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: Tresiba
  Arms: Afrezza + Insulin Degludec
Device: Continuous Subcutaneous Insulin Infusion (CSII) pump with Automatic Insulin Delivery (AID) — Acceptable AID systems in this study are Medtronic 670G/770G and Tandem Control IQ
  Arms: AID Control; Afrezza + Automatic Insulin Delivery

SUMMARY:
A phase 4 study evaluating the efficacy of mealtime control with Afrezza in combination with an automated insulin pump or insulin degludec in adult subjects with type 1 diabetes

DETAILED DESCRIPTION:
MKC-TI-192 is a Phase 4, 90-day, randomized, three-arm, multicenter clinical trial evaluating the treatment paradigm and efficacy of Afrezza in controlling postprandial glucose in adult subjects (≥18 years of age) with Type 1 Diabetes Mellitus (T1DM). Subjects will be randomized to one of three treatment groups (two Afrezza groups and one control group):

* Afrezza + AID: Subjects in this group will use Afrezza for their bolus (mealtime) insulin and a continuous subcutaneous insulin infusion (CSII) pump with an automatic insulin delivery (AID) algorithm using rapid acting analogs (RAA) for their basal and correction insulin coverage.
* Afrezza + Insulin Degludec: Subjects in this group will use Afrezza for their bolus (mealtime and correction) insulin and insulin degludec for basal insulin coverage.
* AID Control: Subjects in this group will use a CSII pump with an AID algorithm using RAA for all bolus (mealtime and correction) and basal insulin coverage (control group).

The study is composed of up to 5 clinic visits (screening, 3 treatment visits, and an end-of-treatment visit) and 9 telephone visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age at the time of signing the informed consent form
* Clinical diagnosis of Type 1 Diabetes
* HbA1c ≥7.0% and <11.0%
* Treatment with a CSII pump with an AID algorithm (Medtronic 670G/770G or Tandem Control IQ) for at least 3 months
* Ability to pay for their own RAA used in the insulin pump or injections, either through co-pay or self-pay, for the duration of the study
* Willingness to follow study procedures including discontinuing their insulin pump and transitioning to insulin degludec injections plus Afrezza

Exclusion Criteria:

* A recent history of asthma (defined as using any medications to treat within the last year), chronic obstructive pulmonary disease (COPD), or any other clinically important pulmonary disease (e.g., cystic fibrosis, bronchopulmonary dysplasia), or significant congenital or acquired cardiopulmonary disease
* History of serious complications of diabetes (e.g., active proliferative retinopathy or symptomatic autonomic neuropathy)
* History of hypersensitivity to insulin or any of the Afrezza excipients
* On dialysis
* Respiratory tract infection within 14 days before screening (subject may return 14 days after resolution of symptoms for rescreening)
* Exposure to any investigational drug in the past 30 days or an investigational device in the past 2 weeks
* Adrenal insufficiency, active use of steroids or planned steroid use
* Hypothyroidism not controlled, as defined by thyroid stimulating hormone (TSH) outside the upper limit of the reference range by >1.5 × in the last 6 months, according to the local laboratory reference range
* Hyperthyroidism not controlled, as defined by TSH below the normal reference range, according to the local laboratory
* Use of antiadrenergic drugs (e.g., beta blockers and clonidine)
* Any concurrent illness (other than diabetes mellitus) not controlled by a stable therapeutic regimen
* History of a significant eating disorder (e.g., anorexia or bulimia nervosa)
* Current drug or alcohol abuse or a history of drug or alcohol abuse that, in the opinion of the Investigator or the Sponsor, would make the subject an unsuitable candidate for participation in the study
* History of smoking (includes cigarettes, cigars, pipes, vaping devices, and marijuana) in the 6 months before screening
* Female subject who is pregnant, breast-feeding, intends to become pregnant, or is of child-bearing potential and not using adequate contraceptive methods as required by local regulation or practice (may include sexual abstinence)
* An event of severe hypoglycemia, as reported by the patient, within the last 180 days before screening
* An episode of diabetic ketoacidosis (DKA), as determined by the Investigator, requiring hospitalization within the last 180 days before screening
* Exposure to Afrezza in the 30 days before screening
* Abnormal TSH or creatinine levels above 2.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kaiserman, MD, Study Director — Mannkind Corporation
Locations (2):
- United States (2):
  - Diabetes Treatment Center, Loma Linda University, Loma Linda, California
  - Texas Diabetes and Endocrinology, Austin, Texas

REFERENCES:
- [Derived] Jacobson C, Kaiserman KB, Ulloa J, Pleitez J, Sylvan J, Rinker J, Codorniz K, Lee S, Vakhshoori M, Lobo Moreno P, Blevins T. Safety and Efficacy of Inhaled Technosphere(R) Insulin in the Postprandial Period With Modified Initial Dose Conversion. Diabetes Ther. 2025 Aug;16(8):1695-1705. doi: 10.1007/s13300-025-01760-5. Epub 2025 Jun 18. PMID 40531276

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, participants who complete the informed consent process are enrolled in the study. In this study, 33 participants were enrolled in the study. The study has a run-in period of up to 28 days. After completion of the run-in period, and confirmation of all eligibility requirements, the participant may be assigned to a study arm/group. In this study, only 28 participants started the treatment phase and were assigned to a study arm/group (5 participants are considered PreRand drops).
Groups:
- Afrezza + Automatic Insulin Delivery (AID): Subjects in this group will use Afrezza for their bolus (mealtime) insulin and a Continuous Subcutaneous Insulin Infusion (CSII) pump with an AID algorithm using Rapid Acting Insulin Analogs (RAA) for their basal and correction insulin coverage.
  Afrezza (insulin human) Inhalation Powder: Pharmaceutical form: powder
  Route of administration: inhalation
  CSII pump with AID: Acceptable AID systems in this study are Medtronic 670G/770G and Tandem Control IQ
- Afrezza + Insulin Degludec: Subjects in this group will use Afrezza for their bolus (mealtime and correction) insulin and insulin degludec for basal insulin coverage.
  Afrezza (insulin human) Inhalation Powder: Pharmaceutical form: powder
  Route of administration: inhalation
  insulin degludec: Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
- AID Control: Subjects in this group will use a CSII pump with an AID algorithm using RAA for all bolus (mealtime and correction) and basal insulin coverage (control group).
  CSII pump with AID: Acceptable AID systems in this study are Medtronic 670G/770G and Tandem Control IQ
Period: Overall Study
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Started | 13 | 10 | 5
Completed | 9 | 10 | 5
Not Completed | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control | Total
Number analyzed (Participants) | 13 | 10 | 5 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 5 | 28
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 3 | 19
  Male | 6 | 1 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 10 | 10 | 5 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 10 | 5 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change in glycated hemoglobin (HbA1c) from baseline to end of study
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percent of glycated hemoglobin
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 9 | 10 | 5
percent of glycated hemoglobin | 0.32 (0.55) | 0.35 (0.58) | 0.52 (0.29)

2. Secondary Outcome: Events of Level 1 Hypoglycemia (SMBG < 70mg/dL)
Description: Events of hypoglycemia (SMBG <70 mg/dL for SMBG values more than 30 minutes apart)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Count of events
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 11 | 10 | 5
Count of events | 12 (12) | 20 (12) | 14 (7)

3. Secondary Outcome: Events of Level 2 Hypoglycemia (SMBG < 54 mg/dL)
Description: Events of hypoglycemia (SMBG <54 mg/dL for SMBG values more than 30 minutes apart)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Count of events
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 11 | 10 | 5
Count of events | 3 (3) | 5 (4) | 4 (5)

4. Secondary Outcome: Events of Severe Hypoglycemia
Description: Events of severe hypoglycemia requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions
Time Frame: 90 days
Measure: Number; unit: Count of events
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 11 | 10 | 5
Count of events | 0 | 0 | 0

5. Secondary Outcome: Change in Time in Range (Glucose of 70 - 180 mg/dL)
Description: Change from baseline to end of study in Time in Range (TIR), defined as the percentage of time spent with glucose in the range of 70 to 180 mg/dL, based on continuous glucose monitoring derived glucose values
Time Frame: baseline and 90 days
Measure: Mean (Standard Deviation); unit: percent of TIR
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 9 | 10 | 5
percent of TIR | 4.69 (27.61) | -3.89 (16.00) | 1.99 (10.12)

6. Secondary Outcome: Change in Time Below Range (Glucose <70 mg/dL)
Description: Change from baseline to end of study in Time Below Range (TBR), defined as the percentage of time spent with glucose <70 mg/dL, based on continuous glucose monitoring derived glucose values
Time Frame: baseline and 90 days
Measure: Mean (Standard Deviation); unit: percent of TBR
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 9 | 10 | 5
percent of TBR | -0.06 (1.72) | 1.92 (4.23) | -0.18 (0.44)

7. Secondary Outcome: Change in Percentage of Time With Glucose <54 mg/dL
Description: Change from baseline to end of study in percentage of time spent with glucose <54 mg/dL, based on continuous glucose monitoring derived glucose values
Time Frame: baseline and 90 days
Measure: Mean (Standard Deviation); unit: percent of time with glucose <54mg/dL
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 9 | 10 | 5
percent of time with glucose <54mg/dL | 0.03 (0.43) | 0.88 (2.04) | -0.1 (0.12)

8. Secondary Outcome: Change in Time Above Range (Glucose >180 mg/dL)
Description: Change from baseline to end of study in Time Above Range (TAR), defined as the percentage of time spent with glucose >180 mg/dL, based on continuous glucose monitoring derived glucose values
Time Frame: baseline and 90 days
Measure: Mean (Standard Deviation); unit: percent of TAR
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 9 | 10 | 5
percent of TAR | -4.63 (28.69) | 1.97 (17.89) | -1.81 (10.17)

9. Secondary Outcome: Change in Percentage of Time With Glucose >250 mg/dL
Description: Change from baseline to end of study in percentage of time spent with glucose >250 mg/dL, based on continuous glucose monitoring derived glucose values
Time Frame: baseline and 90 days
Measure: Mean (Standard Deviation); unit: percent of time with glucose >250mg/dL
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 9 | 10 | 5
percent of time with glucose >250mg/dL | -1.04 (23.57) | 0.84 (9.86) | -4.47 (3.03)

10. Secondary Outcome: Change in Coefficient of Variation (CV)
Description: Change from baseline to end of study in glycemic variability as measured by coefficient of variation (CV), based on continuous glucose monitoring derived glucose values
Time Frame: baseline and 90 days
Measure: Mean (Standard Deviation); unit: percent of coefficient of variation
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 9 | 10 | 5
percent of coefficient of variation | 1 (5) | 4 (9) | -5 (3)

11. Other Pre Specified Outcome: Change in Percent Predicted Forced Expiratory Volume in 1 Second
Description: Change in percent predicted forced expiratory volume in 1 second (FEV1) from baseline to end of study
Time Frame: baseline and 90 days
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 9 | 10 | 5
percent predicted FEV1 | -2 (5) | 2 (6) | -2 (6)

12. Other Pre Specified Outcome: Total Number of Treatment-Emergent Adverse Events
Description: Total Number of Treatment-Emergent Adverse Events (TEAEs)
Time Frame: 90 days
Measure: Number; unit: count of TEAEs
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 13 | 10 | 5
count of TEAEs | 26 | 12 | 1

13. Other Pre Specified Outcome: Total Number of Serious Adverse Events
Description: Total Number of Serious Adverse Events (SAEs)
Time Frame: 90 days
Measure: Number; unit: count of SAEs
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 13 | 10 | 5
count of SAEs | 2 | 1 | 0

14. Other Pre Specified Outcome: Total Number of Adverse Events of Special Interest
Description: Total Number of Adverse Events of Special Interest (AESIs)
Time Frame: 90 days
Measure: Number; unit: count of AESIs
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 13 | 10 | 5
count of AESIs | 3 | 0 | 0

15. Other Pre Specified Outcome: Total Number of Device Complaints
Description: Total Number of Device Complaints
Time Frame: 90 days
Measure: Number; unit: Count of Device Complaints
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
Number analyzed (Participants) | 13 | 10 | 5
Count of Device Complaints | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected for a period of up to 120 days.
Arm/Group | Afrezza + Automatic Insulin Delivery (AID) | Afrezza + Insulin Degludec | AID Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/10 | 0/5
Other Adverse Events (participants affected / at risk) | 7/13 | 8/10 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afrezza + Automatic Insulin Delivery (AID) (N=13) | Afrezza + Insulin Degludec (N=10) | AID Control (N=5)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afrezza + Automatic Insulin Delivery (AID) (N=13) | Afrezza + Insulin Degludec (N=10) | AID Control (N=5)
COVID-19 respiratory infection (Infections and infestations) | 4 (5) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Secondary to COVID19
Decreased Appetitie (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Respiration Abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of the study include its open-label and non-controlled study design and a small sample size (Total Started=28).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the Institution nor the Principal Investigator will disclose any of the results arising out of or in connection with the Clinical Trial or information provided by the Sponsor to the Institution without the prior express written consent of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT05243628/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT05243628/SAP_001.pdf